CLINICAL TRIAL: NCT02997631
Title: A Randomized Controlled Trial of Humanoid Robot-Based Distraction for Venipuncture Pain: The MEDi Study
Brief Title: Robot-Based Distraction to Reduce Pain and Distress in the Pediatric Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00068199
Record Dates: First submitted 2016-12-13; First posted 2016-12-20 (Estimated); Last update posted 2024-09-19 (Actual); Status verified 2018-05

CONDITIONS: Children Requiring IV Placement
Keywords: Pain Management; Distraction Therapy; Robot Based Distraction; MEDi
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MEDi Distraction (Experimental): The intervention will be the use of the MEDi robot. The robot will be at the child's eye level, and will be programmed to introduce itself, interact with the child, and make encouraging comments about how brave he/she was. The duration of its actions will coincide with the length of the procedure (approximately 5-8 minutes).
  Interventions: Device: MEDi Robot
- Standard Care (No Intervention): The control group will receive standard care, which generally includes the use of topical anesthetic cream. This comparison is based on the pragmatic preferences of physicians at the Stollery Children's Hospital as well as precedent in the literature. Overall, it is felt that any new intervention (e.g., the MEDi robot) should be compared to what is currently in practice (i.e., standard care), as no single distraction therapy is consistently and routinely employed in EDs at this time.

INTERVENTIONS:
Device: MEDi Robot — Distraction therapy using an interactive humanoid robot
  Arms: MEDi Distraction

SUMMARY:
Intravenous (IV) insertion is one of the most common procedures for children seeking medical treatment in the Emergency Department (ED). This procedure is often painful and distressing for children and families. This can result in an uncooperative child, a need for multiple cannulation attempts, needle phobia, and dissatisfaction with care for family and healthcare workers. Non-pharmacological treatments are emerging as a newly favoured adjunct to pharmacotherapy, such as distraction therapy.

Distraction therapy involves engaging children in cognitive tasks in order to divert attention from painful stimuli and reduce pain and distress. Currently, distraction therapy is not utilized as a standard of care in the ED. Given children's enthusiasm for technological devices, we propose that the use of a technologically enhanced device may be a more effective distractor and may have a greater impact on pain reduction outcomes of patient importance. The primary objective of this study is to compare the reduction of pain and distress with the use of distraction (via the MEDi robot) versus current standard care in children aged 6 to 11 years who are undergoing IV placement.

DETAILED DESCRIPTION:
Setting and Study Period: This study is a randomized controlled trial and will be conducted in the Emergency Department of the Stollery Children's Hospital (SCH). The SCH is a tertiary care hospital in Edmonton, Alberta whose annual ED census is >50,000 children. Based on our team's previous successful work in this field,12 months of patient recruitment is anticipated, and projected to occur from February 2017 to January 2018.

Study Population: The study will include children aged 6-11 years attending the SCH ED, and requiring an IV placement. See Eligibility section for detailed inclusion/ exclusion criteria. We plan to recruit 80 patients, overall.

Recruitment: Research Assistants (RAs) will be on shift from approximately 15:00 to 23:00 seven days a week. This time corresponds with peak visits requiring IV placements based on data collected from previous studies conducted in the SCH ED. RAs will identify and approach patients aged 6-11 years who require an IV placement. Inclusion/ exclusion criteria will be further assessed, and if the child is eligible, the RA will explain the study and invite the parent and child to participate. After obtaining written, informed consent from the parent (and assent from the child, if applicable), the RA will randomize the patient into one of two study arms and begin data collection. The RA will ask one parent/ caregiver for each child to participate and complete all relevant questionnaires.

Study Assessments: After consent/ assent has been obtained, the RA will collect information from the parent on baseline demographic variables (ex. age, gender), presenting signs and symptoms (ex. chief complaint), as well as previous history with ED visits and IV placement. Before the procedure, the RA will bring the MEDi (Medicine and Engineering Designing intelligence) robot into the room for children in the distraction group, set it up, and explain how to interact with it. The staff nurse will then perform the routine set up for IV placement. Pain will be measured using the child's self-reported scores on the Faces Pain Scale Revised (FPS-R). These scores will be collected immediately before and after IV placement has occurred. The child's response behaviors to pain will be assessed using the Observational Scale of Behavioral Distress (OSBD). The procedure and child will be video-taped during IV insertion to complete the OSBD scoring. Parental anxiety will be measured pre and post procedure with the State Trait Anxiety Inventory - State Scale Revised Version (STAI-S, Form Y). The degree of the child's engagement with the robot will be measured immediately following the procedure with the Intrinsic Motivation Inventory (IMI). Additionally, vitals will be collected pre, post and during the procedure. Data will be entered in real-time into a secure online database hosted on REDCap (Research Electronic Data Capture).

Randomization, Allocation and Blinding of Study Treatment: Randomization will be determined using a secure online randomization tool, through REDCap, and hosted via the Clinical Research Informatics Core at the University of Alberta. A trained RA will obtain the computer-generated randomized assignment after child and parent consent/assent has been obtained. Allocation will be concealed from the research staff, ED staff, and participants until after consent and randomization has been assigned by computer. Due to the nature of the intervention, it will not be possible to blind the children, parents, RAs, or ED staff. The children and their parents will be informed that the study is to evaluate different forms of distraction but will not know the study hypothesis for the MEDi robot. The data analyst will be blind to treatment assignment through the use of randomization codes that will not identify groups until analysis is complete.

Study Intervention and Comparison: The intervention will be the use of the MEDi robot. The robot will be at the child's eye level, and will be programmed to introduce itself, interact with the child, and make encouraging comments about how brave he/she was. The duration of its actions will coincide with the length of the procedure (approximately 5-8 minutes). The control group will receive standard care, which generally includes the use of topical anesthetic cream. This comparison is based on the pragmatic preferences of physicians at the Stollery Children's Hospital as well as precedent in the literature.Overall, it is felt that any new intervention (e.g., the MEDi robot) should be compared to what is currently in practice (i.e., standard care), as no single distraction therapy is consistently and routinely employed in EDs at this time.

ELIGIBILITY:
Inclusion Criteria:

* 6 to 11 years of age
* Needs an IV placement
* Fully conscious and alert
* Has sufficient knowledge of the English language to understand and complete the pain assessments
* Accompanied by a legal guardian.

Exclusion Criteria:

* Hearing or visual impairments
* Neurocognitive delays
* Sensory impairment to pain (e.g., spina bifida)
* Previous enrollment in the same study
* Other exclusion at the discretion of the clinical staff

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 86 (Actual)
Dates: Start 2017-04-20 (Actual); Primary Completion 2018-05-13 (Actual); Study Completion 2018-05-13 (Actual)

PRIMARY OUTCOMES:
Pain of IV insertion | <5 minutes before IV placement, and immediately after IV placement
  Pain scores will be self-reported by the child on the Faces Pain Scale-Revised (FPS-R)
Distress associated with IV insertion | During continuous 15-second intervals before, during, and after the IV placement procedure. Approximately 5 minutes before and after the procedure will be captured.
  Two RAs will independently observe a videotape of each child and use the Observational Scale of Behavioral Distress (OSBD) to assess children's response behaviors to pain.

SECONDARY OUTCOMES:
Parental anxiety | Immediately before and after IV placement
  Measured with the State Trait Anxiety Inventory - State Scale Revised Version (STAI-S, Form Y), a validated and commonly used version of STAI, which has improved psychometric properties
Degree of child's engagement with robot | Approximately 2-5 minutes after IV placement
  To determine a child's degree of engagement with the robotic technology, children, parents, and nurses will complete the 18-item version of the Intrinsic Motivation Inventory

CONTACTS AND LOCATIONS:
Overall Officials: Samina Ali, MD, Principal Investigator — University of Alberta/Stollery Children's Hospital
Locations (1):
- Stollery Children's Hospital Emergency Department, Edmonton, Alberta, Canada

REFERENCES:
- [Derived] Ali S, Manaloor R, Ma K, Sivakumar M, Beran T, Scott SD, Vandermeer B, Beirnes N, Graham TAD, Curtis S, Jou H, Hartling L. A randomized trial of robot-based distraction to reduce children's distress and pain during intravenous insertion in the emergency department. CJEM. 2021 Jan;23(1):85-93. doi: 10.1007/s43678-020-00023-5. Epub 2020 Dec 10. PMID 33683608
- [Derived] Ali S, Sivakumar M, Beran T, Scott SD, Vandermeer B, Curtis S, Jou H, Hartling L. Study protocol for a randomised controlled trial of humanoid robot-based distraction for venipuncture pain in children. BMJ Open. 2018 Dec 14;8(12):e023366. doi: 10.1136/bmjopen-2018-023366. PMID 30552264